CLINICAL TRIAL: NCT05721105
Title: Evaluation of Long-term Quality of Life in Children Supported with ExtraCorporeal Membrane Oxygenation (ECMO): a Prospective Transversal Study
Brief Title: Evaluation of Long-term Quality of Life in Children Supported with ExtraCorporeal Membrane Oxygenation (ECMO)
Acronym: ECMOQoL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0013
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Critical Care
Keywords: Pediatric Intensive Care; Quality of life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ECMO: 50 Patients admitted to pediatric intensive care at the University Hospital of Nantes between January 2014 and December 2022 and supported by ECMO during their hospitalization.
  Interventions: Other: Quality of life assessment using questionnaires
- Control: 50 patients hospitalized at the same age, during the same time period, and sharing the same diagnostic categories as the ECMO group, but the control group never had ECMO.
  Interventions: Other: Quality of life assessment using questionnaires

INTERVENTIONS:
Other: Quality of life assessment using questionnaires — Several quality of life questionnaires will be submitted to the patients and their parents. The questionnaires will be adapted to the age of the patients.

SUMMARY:
The main objective of this prospective transversal comparative study is to describe the quality of life of children supported by ECMO. These patients are described in detail at the Nantes University Hospital, in particular the elements of neurological monitoring. These results will be analyzed in reference to a population hospitalized at the same age, in the same period, and sharing the same diagnostic categories.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted in pediatric intensive care at the Nantes University Hospital between January 2014 and December 2022
* Patients less than 10 years old at admission to the intensive care unit,
* Patients older than 2 years at the time of the cross-sectional evaluation
* For the ECMO group: Patients supported by ECMO
* For the control group: Patient intubated-ventilated for more than 48 hours and/or having received amines and/or having received organ support other than ECMO.
* Patient affiliated to the Social Security.
* Patient with parents who do not object to the study

Exclusion Criteria:

* Known genetic pathology or malformative association at the time of admission to the intensive care unit that could lead to severe neurodevelopmental deficits, independently of the medical events that resulted in the admission to the intensive care unit
* Language difficulty that does not allow for complete information and questionnaire collection

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients included (ECMO group) will be patients under 10 years of age treated by ECMO at the University Hospital of Nantes from January 2014 to December 2022 and who have reached the age of 2 years during the study (the hetero-evaluation questionnaires for the primary endpoint being validated from this age).
  The controls will be patients hospitalized at the same age in pediatric intensive care and at the same periods, who have been intubated and ventilated for at least 48 hours, and/or who have received amines and/or who have benefited from organ support other than ECMO (CONTROL group).
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Compare the overall quality of life of children aged 0-10 years supported by ECMO during their intensive care period with a population of children of the same age hospitalized in pediatric intensive care in the same period. | 15 days
  Quality of life evaluated by the total score of the PedsQL (Pediatric Quality of Life InventoryTM), scale from 0 to 4; 4 being the worst outcome.

SECONDARY OUTCOMES:
To compare the different QoL dimensions of children supported by ECMO between 0 and 10 years of age during their intensive care with reference to a population of children of the same age hospitalized in pediatric intensive care during the same period | up to 15 days
  PedsQL (Pediatric Quality of Life Questionnaire) : Physical functioning, emotional functioning, social functioning, academic functioning.
  PedsQL (Pediatric Quality of Life Questionnaire), scale from 0 to 4; 4 being the worst outcome.
To compare the different QoL dimensions of children supported by ECMO between 0 and 10 years of age during their intensive care stay to a reference consisting of healthy children, not hospitalized, studied over the same period and in the same country | up to 15 days
  PedsQL Questionnaire scores of a cohort of healthy children of the same age from the literature.
  PedsQL (Pediatric Quality of Life InventoryTM), scale from 0 to 4; 4 being the worst outcome.
Describe the association between neurological complications and their severity (seizures, clinical deficits, imaging lesions) and QoL in patients supported by ECMO. | up to 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided